CLINICAL TRIAL: NCT01399983
Title: Assessment of Exercise Capacity and Standardization of Six Minute Walk Test in Patients With Pulmonary Hypertension
Brief Title: Standardization of 6 Minute Walk Test
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 23-069 ex 10/11
Record Dates: First submitted 2011-07-12; First posted 2011-07-22 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Pulmonary Hypertension
Keywords: six minute walk
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pulmonary hypertension: patients with pulmonary hypertension and with exercise-induced pulmonary hypertension take part

SUMMARY:
The 6 minute walk (6MW) gives information about the exercise capacity and it is an important tool for clinical decisions and for the prognostic evaluation of PH patients. The test is technically simple to perform, inexpensive and reproducible. During the 6MW O2 saturation, heart rate, walking distance (in this study after every minute) and the level of dyspnea (BORG-dyspnea scale) may be recorded; however, at present, mainly the walking distance is evaluated. The test is sometimes criticized, because of the dependence on the patient's motivation.

The purpose of the present study is to standardize the test by the incorporation of objective factors. The investigators are correlating the change of heart rate and dyspnea (BORG scale) with the achieved walking distance during subsequent examinations performed with different effort.

DETAILED DESCRIPTION:
On two different days the patients have to absolve four 6MW on different levels of effort - on both days a traditional test will be performed and additionally a test with more effort or with less effort. The order of the tests will be randomized. These two days of the examinations should be within a maximum of three months, provided that there is no sign of relevant clinical changes. After every minute the walking distance is determined. Heart rate and the O2 saturation are measured by pulsoxymetry during the whole test. Every two minutes the patients are asked about their dyspnea (Borg scale).

The purpose of the present study is to standardize the test by the incorporation of objective factors and to detect the correlation between the walking distance and the level of effort during exercise. The investigators expect that the reliability and objectivity of 6MW may increase by the standardization.

The additionally performed cardiopulmonary exercise testing helps to evaluate and stratify patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of pulmonary hypertension or exercise-induced pulmonary hypertension by right heart catheterisation
* informed consent

Exclusion Criteria:

* Myocardiac Infarct within the last 12 months
* Uncontrolled ventricular arrhythmia
* Uncontrolled bradycardic or tachycardic supraventricular arrhythmia
* relevant operations within the last 12 weeks
* change of the hemodynamic therapy within the last 6 weeks
* joint diseases or diseases of peripheral vessels and nerves which may make the results of the six minute walk test unreliable

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pulmonary hypertension or exercise-induced pulmonary hypertension assessed by right heart catheterisation
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
change of six minute walk distance between baseline measurement and measurement with more effort or less effort | the six minute walk test with a different effort is performed 1 hour after the baseline test. The second baseline test and the missing test with a different effort takes place within three months.
  distance at six minute walk performed by different efforts

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria